CLINICAL TRIAL: NCT02816034
Title: Alterations in Cerebellar-dependent Adaptation Due to Cannabis Use Measured With an Explicit-implicit Visuo-motor Learning Paradigm
Brief Title: Cerebellar Alterations in Individuals With a Cannabis Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Pompeu Fabra (Other)
Collaborators: Hospital Clinic of Barcelona (Other); Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other)
Responsible Party: Principal Investigator, Paul Verschure, Professor, Universitat Pompeu Fabra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CannabinoidsCerebellum
Record Dates: First submitted 2016-06-06; First posted 2016-06-28 (Estimated); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Cannabis
Keywords: Learning; Cerebellum
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Experimental Explicit (Experimental): Cannabis user performs visuo-motor rotation tasks informed of an explicit strategy to maximise performance
  Interventions: Behavioral: Visuo-motor rotation; Behavioral: Explicit strategy
- Control Explicit (Active Comparator): Healthy subject performs visuo-motor rotation tasks informed of an explicit strategy to maximise performance
  Interventions: Behavioral: Visuo-motor rotation
- Experimental Implicit (Experimental): Cannabis user performs visuo-motor rotation tasks without being informed of the explicit strategy
  Interventions: Behavioral: Visuo-motor rotation; Behavioral: Explicit strategy
- Control Implicit (Active Comparator): Healthy subject performs visuo-motor rotation tasks without being informed of the explicit strategy
  Interventions: Behavioral: Visuo-motor rotation

INTERVENTIONS:
Behavioral: Visuo-motor rotation — Participant moves a cursor on a screen by sliding a pen over a digital tablet. Participants perform a center-out movement, aiming to a target that appears over one of a set of eight markers radially distributed. In several block of trials, the mapping of the pen position to the cursor is rotated.
Behavioral: Explicit strategy — Participant is provided with an explicit instruction as to how counteract the effects of the visuo-motor rotation via aiming to a marker adjacent target
  Arms: Experimental Explicit; Experimental Implicit

SUMMARY:
The purpose of this study is to investigate if individuals with a cannabis use disorder have an impaired cerebellar function by assessing possible alterations to their implicit adaptation during a visuomotor rotation task.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with a Cannabis use disorder following Diagnostic and Statistical Manual (DSM-V) criteria.
* Patients screen positive to cannabis in the urine analysis performed a week prior to assessment.
* Right-handed patients.
* Patients provide a signed consent.

Exclusion Criteria:

* Patients with another current substance use disorder (with the exception of tobacco).
* Patients with a visual impairment that has not been corrected.
* Patients with a cognitive impairment such as mental retardation.
* Patients with psychotic disorders.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Directional error of hand trajectories towards a target | 1 day (a single session)

SECONDARY OUTCOMES:
Reaction times | 1 day (a single session)
Intrinsic Motivational Inventory | 1 day (a single session)

REFERENCES:
- [Background] Taylor JA, Klemfuss NM, Ivry RB. An explicit strategy prevails when the cerebellum fails to compute movement errors. Cerebellum. 2010 Dec;9(4):580-6. doi: 10.1007/s12311-010-0201-x. PMID 20697860
- [Background] Mazzoni P, Krakauer JW. An implicit plan overrides an explicit strategy during visuomotor adaptation. J Neurosci. 2006 Apr 5;26(14):3642-5. doi: 10.1523/JNEUROSCI.5317-05.2006. PMID 16597717